CLINICAL TRIAL: NCT03473600
Title: Cryotherapy Versus Intralesional Corticosteroid Injection In Treatment Of Alopecia Areata: Trichoscopic Evaluation
Brief Title: Cryotherapy Versus Steroids In Alopecia Areata:Trichoscopic Evaluation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noura Ali, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVILCsAA
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Cryotherapy; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): •The first group (20 patients) will be treated with cryotherapy using liquid nitrogen spray, two cycles each one 3-5 seconds, one session every two weeks, for three months.
  Interventions: Procedure: Cryotherapy
- control group (Active Comparator): •The second group (20 patients) will be treated with intralesional injection of 4mg/ml/ session of triamcinolone-acetonide, it will be injected into deep dermis or upper subcutaneous tissue using a 0.5-inch long 30-gauge needle at multiple sites, 1 cm apart and 0.1 ml into each site, once every three weeks, for three months, using insulin syringes.
  Interventions: Drug: Triamcinolone acetonide injection

INTERVENTIONS:
Procedure: Cryotherapy — Liquid Nitrogen spray
  Arms: study group
Drug: Triamcinolone acetonide injection — Intralesional Triamcinolone Acetonide injection
  Arms: control group

SUMMARY:
Alopecia areata is the most frequent cause of inflammation-induced hair loss with prevalence from 0.1 to 0.2%. It has no age nor sex predilection .

Clinically, alopecia areata presents as a well-circumscribed patch of sudden hair loss. It affects any hair bearing area. The most common affected site is the scalp. Based on site and extent, AA can be classified into; diffuse, multi-locularis, mono-locularis, totalis, universalis, and ophiasis.

DETAILED DESCRIPTION:
Histologically, lesional biopsies of alopecia areata demonstrate a peri_follicullare and intra_folliculare mononuclear cell infiltrate around anagen phase hair follicles .The infiltrate consists mostly of activated lymphocytes in particular CD4 cells as well as dendritic cells and macrophages.

Many theories were implicated in pathogenesis of alopecia areata such as; autoimmune lymphocytic attack of the hair, genetic basis and environmental factors. So the pathogenesis of alopecia areata remains to be determined. Currently a widely accepted theory is the autoimmune etiology. Specific T_cell lymphocytes, autoantibodies against anagen follicles, and various cytokines such as interferon-γ, interleukins, and tumor necrosis factor-α have been found to play a major role in alopecia areata. In addition, the immune privilege theory has been recently introduced and suggested to play a role in the pathogenesis.

Many kinds of treatment modalities are present in localized alopecia areata. Injectable forms of corticosteroids are first line of alopecia areata therapy, and also topical use of steroids is widely used. Others are topical sensitization with anthrain, minoxidil and cryotherapy. In extention form of alopecia areata, systemic treatments like corticosteroids, cyclosporine and methotrexate can be used.

Intralesional Corticosteroid injection:

National Guidelines from British Association of Dermatologists, recommend intralesional corticosteroid therapy as the first line treatment for localized patchy alopecia areata, with approximate success rates of 60-75%. Their use was first described in 1958, with the use of hydrocortisone.

Immunosuppression is the main mechanism of action. Corticosteroids suppress the T-cell-mediated immune attack on the hair follicle. Steroids with low solubility are preferred for their slow absorption from the injection site, promoting maximum local action with minimal systemic effect. The efficacy of intralesional corticosteroid injection is variable depending on the patient population treated.

Cryotherapy:

Cryotherapy may act through either singly or by a combination of the following mechanisms resulting in hair regrowth in alopecia areata. After initial vasoconstriction with cryotherapy, there is a significant local vasodilatation during the thaw period as the temperature reaches zero degree Celsius. Thus, cryotherapy is speculated to dilate the vessels around the affected hair follicles, with an increase in the blood flow leading to follicular hair regrowth. Moreover, local edema and inflammation occurring after cryotherapy may play a role in inducing vasodilation.

Cryotherapy is also speculated to inflict partial damage to keratinocytes, especially the antigenic components of the hair follicle keratin16 and trichohyalin, which are targeted by antibodies and thus, further decrease in damaging perifollicular infiltrate.

Cryotherapy may also alter tissue Langerhans cells, which in turn could alter the process of antigen presentation with further decrease in T cell infiltration. As it is known, the white hairs are spared in alopecia areata; it is hypothesized that melanocytes may have a role in the pathogenesis ofalopecia areata. Hence, cryotherapy may also act by destructing the melanocytes further preventing their role in the initiation of alopecia areata.

Dermoscopy:

Dermoscopy is now considered as a valuable tool in diagnosis of variable skin lesions. It is a non-invasive procedure which was initially used to assess pigmented lesions.

Scalp dermoscopy (Trichoscopy) does not only facilitate diagnosis of hair disorders but also give clues about disease stage and progression. Trichoscopy allows the superimposition of the skin layers with the possibility to observe any surface or deep skin layers.

The most common trichoscopic features of alopecia areata are yellow dots, micro-exclamation mark hairs, tapered hairs, black dots, broken hairs, and regrowing upright or regrowing coiled hairs. Black dots as remnants of exclamation mark hairs or broken hairs provide a sensitive marker for disease activity as well as severity of alopecia areata. Yellow dots, are considered to be the most sensitive dermoscopic feature of alopecia areata. Tapering hair is considered as a marker of disease activity and known to reflect exacerbation of disease. Trichoscopic characteristics have a clinical significance in alopecia areata for diagnosis and prognosis.

Severity of alopecia tool Score:

National Alopecia Areata Foundation working committee has devised "Severity of Alopecia Tool score. Severity of alopecia tool score is useful to find out the quantitative assessment of scalp hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Age >12 years.
* Both sexes will be included.
* Newly diagnosed cases.

Exclusion Criteria:

* Children < 12 years.
* Pregnancy and lactation.
* Patients with active scalp infection.
* Patients with cold sensitivity (regarding the first group).
* Any newly onset medical systemic illness.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The incidence of patietns with hair regrowth | 3 months
  measuring severity of alopecia tool score and dermoscopic examination

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alkhalifah A, Alsantali A, Wang E, McElwee KJ, Shapiro J. Alopecia areata update: part I. Clinical picture, histopathology, and pathogenesis. J Am Acad Dermatol. 2010 Feb;62(2):177-88, quiz 189-90. doi: 10.1016/j.jaad.2009.10.032. PMID 20115945
- [Background] Campos-do-Carmo G, Ramos-e-Silva M. Dermoscopy: basic concepts. Int J Dermatol. 2008 Jul;47(7):712-9. doi: 10.1111/j.1365-4632.2008.03556.x. PMID 18613881
- [Background] Chang KH, Rojhirunsakool S, Goldberg LJ. Treatment of severe alopecia areata with intralesional steroid injections. J Drugs Dermatol. 2009 Oct;8(10):909-12. PMID 19852119
- [Background] Gilhar A, Etzioni A, Paus R. Alopecia areata. N Engl J Med. 2012 Apr 19;366(16):1515-25. doi: 10.1056/NEJMra1103442. No abstract available. PMID 22512484
- [Background] Gilhar A, Paus R, Kalish RS. Lymphocytes, neuropeptides, and genes involved in alopecia areata. J Clin Invest. 2007 Aug;117(8):2019-27. doi: 10.1172/JCI31942. PMID 17671634
- [Background] Gregoriou S, Papafragkaki D, Kontochristopoulos G, Rallis E, Kalogeromitros D, Rigopoulos D. Cytokines and other mediators in alopecia areata. Mediators Inflamm. 2010;2010:928030. doi: 10.1155/2010/928030. Epub 2010 Mar 11. PMID 20300578
- [Background] Inui S, Nakajima T, Itami S. Significance of dermoscopy in acute diffuse and total alopecia of the female scalp: review of twenty cases. Dermatology. 2008;217(4):333-6. doi: 10.1159/000155644. Epub 2008 Sep 18. PMID 18799878
- [Background] KALKOFF KW, MACHER E. [Growing of hair in alopecia areata & maligna after intracutaneous hydrocortisone injection]. Hautarzt. 1958 Oct;9(10):441-51. No abstract available. German. PMID 13610145
- [Background] Kang H, Wu WY, Lo BK, Yu M, Leung G, Shapiro J, McElwee KJ. Hair follicles from alopecia areata patients exhibit alterations in immune privilege-associated gene expression in advance of hair loss. J Invest Dermatol. 2010 Nov;130(11):2677-80. doi: 10.1038/jid.2010.180. Epub 2010 Jul 8. No abstract available. PMID 20613773
- [Background] Madani S, Shapiro J. Alopecia areata update. J Am Acad Dermatol. 2000 Apr;42(4):549-66; quiz 567-70. PMID 10727299
- [Background] Mane M, Nath AK, Thappa DM. Utility of dermoscopy in alopecia areata. Indian J Dermatol. 2011 Jul;56(4):407-11. doi: 10.4103/0019-5154.84768. PMID 21965849
- [Background] Olsen EA, Hordinsky MK, Price VH, Roberts JL, Shapiro J, Canfield D, Duvic M, King LE Jr, McMichael AJ, Randall VA, Turner ML, Sperling L, Whiting DA, Norris D; National Alopecia Areata Foundation. Alopecia areata investigational assessment guidelines--Part II. National Alopecia Areata Foundation. J Am Acad Dermatol. 2004 Sep;51(3):440-7. doi: 10.1016/j.jaad.2003.09.032. No abstract available. PMID 15337988
- [Background] Pimentel CB, Moraes AM, Cintra ML. Angiogenic effects of cryosurgery with liquid nitrogen on the normal skin of rats, through morphometric study. An Bras Dermatol. 2014 May-Jun;89(3):410-3. doi: 10.1590/abd1806-4841.20142249. PMID 24937813
- [Background] Rodriguez TA, Duvic M; National Alopecia Areata Registry. Onset of alopecia areata after Epstein-Barr virus infectious mononucleosis. J Am Acad Dermatol. 2008 Jul;59(1):137-9. doi: 10.1016/j.jaad.2008.02.005. Epub 2008 Mar 7. PMID 18329131
- [Background] Rudnicka L, Olszewska M, Rakowska A, Slowinska M. Trichoscopy update 2011. J Dermatol Case Rep. 2011 Dec 12;5(4):82-8. doi: 10.3315/jdcr.2011.1083. PMID 22408709
- [Background] Sawaya ME, Hordinsky MK. Glucocorticoid regulation of hair growth in alopecia areata. J Invest Dermatol. 1995 May;104(5 Suppl):30S. doi: 10.1038/jid.1995.49. No abstract available. PMID 7738385
- [Background] Seetharam KA. Alopecia areata: an update. Indian J Dermatol Venereol Leprol. 2013 Sep-Oct;79(5):563-75. doi: 10.4103/0378-6323.116725. PMID 23974575
- [Background] Shapiro J. Current treatment of alopecia areata. J Investig Dermatol Symp Proc. 2013 Dec;16(1):S42-4. doi: 10.1038/jidsymp.2013.14. PMID 24326551
- [Background] Tosti A, Iorizzo M, Botta GL, Milani M. Efficacy and safety of a new clobetasol propionate 0.05% foam in alopecia areata: a randomized, double-blind placebo-controlled trial. J Eur Acad Dermatol Venereol. 2006 Nov;20(10):1243-7. doi: 10.1111/j.1468-3083.2006.01781.x. PMID 17062039
- [Background] Wasserman D, Guzman-Sanchez DA, Scott K, McMichael A. Alopecia areata. Int J Dermatol. 2007 Feb;46(2):121-31. doi: 10.1111/j.1365-4632.2007.03193.x. PMID 17269961